CLINICAL TRIAL: NCT07138703
Title: The Effect of Mobile Web-based Intervention Programme on Students' Nursing Education Stress and Sleep Quality
Acronym: application
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fidan Balkaya (Other)
Collaborators: Scientific Research Projects Coordination Unit (Ambiguous)
Responsible Party: Sponsor-Investigator, Fidan Balkaya, Research Asistant, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Nursing
Record Dates: First submitted 2025-08-07; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-06

CONDITIONS: MOBILE WEB-BASED INTERVENTION PROGRAM; NURSING EDUCATION STRESS; SLEEP QUALITY
Keywords: Web-based intervention program, nursing student, stress, sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Experimental Group: The participants in this group will be using the mobile application Control Group: The participants in this group will not be using the mobile application
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The participants in this group will be using the mobile application
  Interventions: Behavioral: Mobile based intervention program
- Control Group (No Intervention): The participants in this group will not be using the mobile application

INTERVENTIONS:
Behavioral: Mobile based intervention program — The participants in this group will be using the mobile application
  Arms: Intervention Group

SUMMARY:
Nursing students experience increased stress and sleep problems due to their demanding academic schedules and the pressures of the clinical environment. Therefore, addressing students' needs for stress and sleep management is critical to improving their educational success. A review of the literature reveals that various interventions are being used to reduce stress levels or improve sleep quality for university students. The purpose of this study is to examine the effects of a web-based intervention program on the stress and sleep levels of nursing students.

This study will utilize a pretest-posttest control group experimental design. The study will be conducted with 120 nursing students enrolled at İnönü University Faculty of Nursing from September 2025 to June 2026. Participants will be administered a Personal Information Form, the Perceived Stress Scale, the Nursing Education Scale, and the Pittsburgh Sleep Quality Index, and the experimental and control groups will be monitored via a mobile application for 12 weeks. Descriptive statistics such as percentages, arithmetic mean (x̄), and standard deviation (SD), along with chi-square and independent samples t-tests, repeated measures t-tests, and Cronbach's alpha will be used for research analyses.

The research is unique in terms of its sample size and the intervention it plans to implement. Therefore, it has the potential to be published in respected international scientific journals. Furthermore, if the effectiveness of the application in managing stress and sleep is established, it is anticipated that it could be applied to other adult populations, particularly midwifery students.

ELIGIBILITY:
Inclusion Criteria:

* PUKI total score above 5
* Individuals with internet access
* Owning an Android or iOS phone
* Those who are open to communication and collaboration

Exclusion Criteria:

* Individuals with a psychiatric diagnosis and use of psychiatric medications, according to ASM records,
* who sleep less than four hours a day, who consume more than four cups of coffee a day
* who have hearing or balance problems (orthopedic or neurological) will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
nursing education stress scores | six months
  The scale consists of a total of 32 items and two subscales: "Application Stress" and "Academic Stress." Items 4, 5, 7, 9, 11, 13, 15, 16, 18, 19, 21, 24, 25, 27, 29, and 32 are scored to calculate students' application stress, while items 1, 2, 3, 6, 8, 10, 12, 14, 17, 20, 22, 23, 26, 28, 30, and 31 are scored to calculate students' academic stress. The scale is a four-point Likert-type scale, with each item scored between 0 and 3 ("0" being not stressful at all, "3" being very stressful). The highest score possible from the scale is 96, with higher scores indicating higher educational stress.
sleep quality | six months
  The PSQI consists of seven components (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance/conditions affecting sleep, use of sleep-inducing medications/substances, and daytime dysfunction/sleepiness). 18 questions are included in the scoring when calculating the PSQI. The answers to each are scored between 0 and 3. The total scale score ranges from 0 to 21. A total scale score higher than 5 indicates poor sleep quality.

IPD SHARING:
Plan to Share IPD: No
Due to ethical and legal restrictions, IPD will not be shared